CLINICAL TRIAL: NCT04050839
Title: The Effectiveness of Pain Neuroscience Education in Patients with Fibromyalgia
Brief Title: Pain Neuroscience Education in Patients with Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Principal Investigator, Kutahya Health Sciences University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KutahyaMSUfibro
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2022-03

CONDITIONS: Pain, Chronic; Fibromyalgia
Keywords: pain neuroscience education; patient education
MeSH Terms: conditions — Chronic Pain; Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neuroscience pain education group (Experimental): Pain neuroscience education in addition medical treatment
  Interventions: Other: Pain neuroscience education; Drug: Medical treatment
- Control group (Active Comparator): Medical treatment only
  Interventions: Drug: Medical treatment

INTERVENTIONS:
Other: Pain neuroscience education — A total of 4 NPE (Neuroscience paine education) sessions were held, once each week in addition medical treatment similar to control group. The NPE sessions were conducted by an experienced physiotherapist certified in NPE in face-to-face, group sessions lasting 40-45 minutes. In NPE, the patient is taught about the physiology of pain, central sensitization, representation of the different body regions in the brain, pain-related changes in body perception, and the psychosocial dimensions of pain.
  Arms: Neuroscience pain education group
Drug: Medical treatment — The patients in control group continued taking their regular gabapentin and pregabalin-derivative drug therapy at the same dosage and duration specified by their physicians.

SUMMARY:
Many patients with fibromyalgia have little understanding of their condition, leading to maladaptive pain cognitions and coping strategies. Current research has suggested the use of physiotherapy and rehabilitation in addition to cognitive patient education in the treatment of fibromyalgia syndrome. This study aimed to explore the effectiveness of pain neuroscience education in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* have fibromyalgia as defined by the criteria of the 1990 ACR
* have Turkish as their native language
* between 18 and 65 years of age

Exclusion Criteria:

* Having cognitive impairment
* Receiving psychotherapy
* Illiterate people
* Patients with significant hearing loss

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | Change from Baseline FIQ at 4th weeks
  The FIQ is an assessment and evaluation instrument developed to measure fibromyalgia (FM) patient status, progress and outcomes
Pressure pain thresholds (PPT) | Change from Baseline PPT at 4th weeks
  Pressure pain thresholds in following five points, 7th cervical vertebra, 3th lumbal vertebra, 5th lumbal vertebra, the belly of calf muscles, and 2nd distal interfalangeal joint were measured using a analog pressure algometer(Baseline, USA).
Tinel's Sign | Change from Baseline PPT at 4th weeks
  The Tinel sign is the result of a simple, noninvasive test that checks for nerve problems. The test is positive when a tingling or prickling sensation is felt in the distribution of the Tibial nerve.

SECONDARY OUTCOMES:
Tampa Scale of Kinesiophobia | Change from Baseline PPT at 4th weeks
  The Tampa Scale for Kinesiophobia (TSK) was used for the assessment of kinesiophobia. The TSK is a 17-item questionnaire developed to measure the fear of movement/re-injury.

CONTACTS AND LOCATIONS:
Locations (1):
- KutahyaMSU, Kütahya, Kutahya Health Sciences University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No